CLINICAL TRIAL: NCT01327469
Title: The Efficacy of 5 Anthelmintic Regimes Against T. Trichiura Infections in Schoolchildren in Jimma, Ethiopia
Brief Title: The Efficacy of Five Anthelmintic Regimes Against Trichuris Trichiura Infections in Schoolchildren in Jimma, Ethiopia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: VLIR-UOS Institutional University Cooperation (Unknown)
Responsible Party: Jozef Vercruysse, University Ghent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010/517
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Infection by Trichuris Trichiura
MeSH Terms: conditions — Trichuriasis | interventions — Albendazole; Mebendazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Albendazole 400mg (Experimental): albendazole, 1 x 400mg
  Interventions: Drug: Albendazole 400mg
- Albendazole 2 x 400mg (Experimental): albendazole, 2 x 400mg
  Interventions: Drug: Albendazole, 2 x 400mg
- Mebendazole 500mg (Experimental): mebendazole, 1 x 500mg
  Interventions: Drug: Mebendazole 500mg
- Mebendazole 2 x 500mg (Experimental): mebendazole, 2x 500mg
  Interventions: Drug: Mebendazole 2 x 500mg
- Pyrantel-oxantel + mebendazole (Experimental): pyrantel-oxantel (10mg/kg)+ mebendazole (500mg)
  Interventions: Drug: Pyrantel-oxantel + mebendazole

INTERVENTIONS:
Drug: Albendazole, 2 x 400mg — Albendazole 2 x 400mg
  Arms: Albendazole 2 x 400mg
Drug: Albendazole 400mg — Albendazole 400mg
  Arms: Albendazole 400mg
Drug: Mebendazole 500mg — Mebendazole 500mg
  Arms: Mebendazole 500mg
Drug: Mebendazole 2 x 500mg — Mebendazole 2 x 500mg
  Arms: Mebendazole 2 x 500mg
Drug: Pyrantel-oxantel + mebendazole — Pyrantel-oxantel + mebendazole
  Arms: Pyrantel-oxantel + mebendazole

SUMMARY:
The major soil-transmitted helminths (STHs), Ascaris lumbricoides (roundworm), Trichuris trichiura (whipworm) and Necator americanus/Ancylostoma duodenal (hookworms) are amongst the most prevalent parasites worldwide. An estimated 4.5 billion individuals are at risk for STH and more than one billion individuals are thought to be infected, of which 450 million have significant morbidity attributable from their infection, school-aged children in particular. In this population infections cause stunting of the linear growth, anemia, reduce the cognitive function and contribute to the existing malnutrition. In Jimma (Ethiopia), STH are highly prevalent, affecting more than 60% of the children (data not published).

Current efforts to control STH infections involve periodic mass drug anthelmintic treatment of infected children in endemic areas and are likely to intensify as more attention is addressed to the importance of these neglected diseases. Monitoring drug efficacy in these control programs has become indispensable in order to detect the emergence of resistance and/or identify confounding factors affecting the drug efficacy. Recently a study has evaluated a single dose albendazole (ALB) in school age children across 7 countries, including Ethiopia, revealing that this regime is highly efficacious for the treatment of A. lumbricoides (99.5%) and hookworms (94.8%), but not for T. trichiura (50.8%). For this parasite a repeated dose regime of ALB on consecutive days is likely to be more appropriate. Alternative drugs are mebendazole (single dose 500mg) and pyrantel+oxantel (single dose 10mg/kg), of which the latter holds promise as it can also be administrated to children between 6 months and 2 years. The main objective of the present study, therefore, is to assess the efficacy of 5 different treatment regimes against T. trichiura in schoolchildren in Jimma, Ethiopia, including albendazole (1 x 400mg, 2 x 400mg), mebendazole (1 x 500mg, 2x 500mg) and pyrantel-oxantel (10mg/kg)+mebendazole (500mg).

ELIGIBILITY:
Inclusion Criteria:

* all school age children who are eligible to participate in the study

Exclusion Criteria:

* Not willing to participate (no informed consent)
* Unable to give samples for follow up
* Severe intercurrent medical condition
* Diarrhea at first sampling
* Study subjects who had treatment for STH in the last 3 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2250 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Efficacy against T. trichiura of various treatment regimes | After two weeks treatment
  The evaluation of the efficacy against T. trichiura of various treatment regimes. To this end, subjects infected with T. trichura (based on McMaster), will be randomly assigned to one of the five proposed treatment regimes. Two weeks after the treatment, faecal egg counts will be performed and the reduction in faecal egg counts will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Vercruysse, PhD, Principal Investigator — University Ghent
Locations (1):
- Jimma University, Jimma, Ethiopia

REFERENCES:
- [Derived] Levecke B, Mekonnen Z, Albonico M, Vercruysse J. The impact of baseline faecal egg counts on the efficacy of single-dose albendazole against Trichuris trichiura. Trans R Soc Trop Med Hyg. 2012 Feb;106(2):128-30. doi: 10.1016/j.trstmh.2011.09.007. Epub 2011 Dec 19. PMID 22189084